CLINICAL TRIAL: NCT02496819
Title: Metacognitive Self-regulated Learning and Sensory Integrative Approaches for Children With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Sydney (Other)
Collaborators: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Karen Liu, Associate Professor, University of Western Sydney
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SR-Autism
Record Dates: First submitted 2015-06-26; First posted 2015-07-14 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Children
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metacognitive self-regulated learning intervention (Experimental): It involves training of daily tasks using a self-correct strategy. Participants' performance will be video-taped and they will then watch the video playback for reflection and self-correction under the guidance of the occupational therapist.
  Interventions: Other: Meta-cognitive self-regulated learning intervention
- Sensory Integration intervention (Experimental): It involves active, fun physical activity completing 8 stations of activities involving tactile, proprioceptive and vestibular tasks. Frequent breaks will be given to avoid exhaustion and fatigue throughout the activities.
  Interventions: Other: Sensory integration intervention
- Activity-Based Intervention (Active Comparator): It provides constructional, drawing and crafts activity. Participants are guided to complete these tasks
  Interventions: Other: Activity-based intervention

INTERVENTIONS:
Other: Meta-cognitive self-regulated learning intervention — It is a 12-week intervention programme with one 60 minutes sessions per week.
  Arms: Metacognitive self-regulated learning intervention
Other: Sensory integration intervention — It is a 12-week intervention programme with one 60 minutes sessions per week.
  Arms: Sensory Integration intervention
Other: Activity-based intervention — It is a 12-week intervention programme with one 60 minutes sessions per week.
  Arms: Activity-Based Intervention

SUMMARY:
Children with Autism Spectrum Disorder (ASD) are increasing each year. There are about 1 in 160 children for the age group of 6-12 years old in Australia are diagnosed with ASD. Children with ASD have impairment in two common areas including: i) social and communication and ii) repetitive and stereotypical patterns of behaviours. These common features result in behavioural problems which negatively impact children's participation in school, activities of daily living and social engagement.

Therefore, there is a need for effective interventions to overcome the behavioural problems in children with ASD.

The purpose of the study is to investigate the effect of sensory integration (SI) and self-regulated learning versus an activity-based control programme in reducing behavioural problems in children with ASD that interfere with their daily livings, school, and social engagement.

The study will adopt a randomized controlled trial design with three intervention groups: I) self-regulated learning, II) sensory integration and III) activity-based intervention as the control group.

DETAILED DESCRIPTION:
Children with Autism Spectrum Disorder (ASD) are commonly associated with behavioural problems which may negatively impact on their participation in school, activities of daily livings and social engagement. In order to minimise the impact on the daily functioning of these children, overcoming the behavioural problems in these children is essential.

Two intervention approaches will be used in this study. These are i) self-regulated learning and ii) sensory integration. Sensory integration is commonly used for children with developmental problems. Self-regulated learning has been used to promote children's self-directed learning and in people with brain injuries.

However, the evidence towards the effectiveness of these two interventions in alleviating the effects of behavioural problems on participation in school, daily and social activities for children with ASD is limited and inconclusive.

Self-regulated learning theory:

The origin of self-regulated learning approach came from Albert Bandura's social cognitive theory. The theory states that intervention affects one's learning by modifying the personal, environmental and behavioural factors. The personal factor refers to one's beliefs and attitudes. The environment factor comprises of feedback, instructions, information gathered from teachers or instructors and also from the assistance of parents and peers. The behavioural factor includes past performance that are socially unacceptable. The key of self-regulated learning is to ensure that children make use of a cognitive strategy to facilitate behaviour learning by helping them to bring problems and solutions towards own consciousness. Several studies had used self-regulated learning in children and adults population. It was found a significant improvement in task performance for children with Attention Deficit Hyperactive Disorders (ADHD). The positive effect was also shown in another study showing improvements in performance measures of reading and intelligence quotient among children with moderate learning disabilities. Similar results were also seen in adults with brain injury in various studies. They suggested that self-regulated learning could enhance the active learning of participants.

Children with ASD were reported to commonly associate with self-regulation problems affecting their behaviour and learning ability. However, there is no study using self-regulated learning for this group of children to alleviate the effect of behavioural problems on their school, daily and social participation.

Sensory integration intervention theory:

Sensory integration theory was developed in 1960s and 1970s. The theory was developed to target on the neurological processing of sensory information. The theory suggests that purposeful behaviours may be interrupted when there is an interference of neurological processing and integration of sensory information. Sensory integration interventions have been widely used in varieties of settings among children with development problems. However, despite the vast amount of literature that exists on the effectiveness of sensory integration intervention, the overall evidence on the effectiveness on children with ASD and behavioural problems remains inconclusive. Some studies showed that sensory integration was an effective intervention given a positive result, but others showed no benefit or inconclusive findings.

Studies previously used sensory integration intervention seemed not using the fidelity measures in the intervention design to ensure that the intervention met the requirement of sensory integration theory. This could be one of the reasons for the inconclusive finding made on its effectiveness. Furthermore, most of the studies used a single-case study design with small sample sizes. In addition, previous studies using sensory integration did not focus on alleviating the effects of behavioural problems on function in the daily livings, school and social engagement for children with ASD.

This study, will therefore, adopt a randomised controlled trial (RCT) design to investigate the effect of sensory integration and self-regulated learning interventions (comparing with activity-based control intervention) in reducing the effects of behavioural problems on daily living, school and social engagement in children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ASD meeting the requirements of the Diagnostic and Statistical Manual of Mental Disorders without dual diagnoses such as physical disabilities
* Overall score ≥ 70 in Part I and Part II of the Vineland Adaptive Behaviour Scales (VABS-II) (2nd ed.). These parts of the scale will assess:.

  * Problem behaviours Part I (internalizing, externalizing, other behaviours): 36 items
  * Problem behaviours Part II (critical items): 14 items
* Have an IQ greater than 50. This is indicative of a normal intelligence quotient (IQ) to moderate grade intellectual disability. This is required so they are able to follow verbal instructions.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Adaptive behaviour on the Vineland Adaptive Behaviour Scales - change from baseline after the intervention | Baseline and after the intervention (12 weeks)
Adaptive behaviour on the Vineland Adaptive Behaviour Scales - change from baseline at one month after the intervention completed | Baseline and one month after the intervention completed (16 weeks)
Executive function behaviours on the Behaviour Rating Inventory of Executive Function - change from baseline after the intervention | Baseline and after the intervention (12 weeks)
Executive function behaviours on the Behaviour Rating Inventory of Executive Function - change from baseline at one month after the intervention completed | Baseline and one month after the intervention completed (16 weeks)
School-related task performance on the School Function Assessment - change from baseline after the intervention | Baseline and after the intervention (12 weeks)
School-related task performance on the School Function Assessment - change from baseline at one month after the intervention completed | Baseline and one month after the intervention completed (16 weeks)
Social skills on the Walker Mc-Connell scale - change from baseline after the intervention | Baseline and after the intervention (12 weeks)
Social skills on the Walker Mc-Connell scale - change from baseline at one month after the intervention completed | Baseline and one month after the intervention completed (16 weeks)

SECONDARY OUTCOMES:
Sensory processing difficulties on the Sensory Processing Measures - change from baseline after the intervention | Baseline and after the intervention (12 weeks)
Sensory processing difficulties on the Sensory Processing Measures - change from baseline at one month after the intervention completed | Baseline and one month after the intervention completed (16 weeks)
Sensory processing patterns and effects on functional performance on the Sensory Profile - change from baseline after the intervention | Baseline and after the intervention (12 weeks)
Sensory processing patterns and effects on functional performance on the Sensory Profile - change from baseline at one month after the intervention completed | Baseline and one month after the intervention completed (16 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Karen P.Y. Liu, PhD, Principal Investigator — Western Sydney University
Locations (1):
- National University of Malaysia, Bangi, Selango, Malaysia

IPD SHARING:
Plan to Share IPD: No